CLINICAL TRIAL: NCT01088269
Title: Evaluation of the Oscillometric Blood Pressure Measurement in Atrial Fibrillation and Relation of Blood Pressure With Serum Biomarkers and Echocardiographic Indexes
Brief Title: Blood Pressure Assessment in Atrial Fibrillation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Athens (Other)
Responsible Party: Principal Investigator, George S. Stergiou, Associate Professor of Medicine and Hypertension, University of Athens
Other Study IDs: BPM IN AF
Record Dates: First submitted 2010-03-16; First posted 2010-03-17 (Estimated); Last update posted 2017-09-14 (Actual); Status verified 2017-09

CONDITIONS: Atrial Fibrillation
Keywords: Blood Pressure Measurement; Atrial Fibrillation; Blood pressure measurement in atrial fibrillation; Atrial Fibrillation diagnosis
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- AF: Hypertensive patients in AF
- Non-AF: Hypertensive Patients

SUMMARY:
This is a cross-sectional study including patients with permanent atrial fibrillation. Assessment will include:

* clinic blood pressure measurements (mercury sphygmomanometer and automated oscillometric device)
* 24-hour ambulatory blood pressure monitoring
* determination of various serum markers and cardiac ultrasound.
* evaluation of a 24h ambulatory blood pressure monitoring device (Microlife WatchBPO3) in terms of its diagnostic value for the detection of atrial fibrillation compared with the reference 24h Holter ECG

ELIGIBILITY:
Inclusion Criteria:

* Hypertensives adults in atrial fibrillation

Exclusion Criteria:

* Renal disease (Cr > 2 mg/l).
* Patients with pacemaker rhythm during the study.
* Each patient with acute disease (inflammation, surgery), malignancy, collagen diseases, pulmonary fibrosis, renal failure, liver failure, chronic inflammatory diseases.

Ages: 25 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: SUBJECTS REFERRED TO HYPERTENSION CENTER
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2010-03; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Blood Pressure Measurement in Atrial Fibrillation,Serum Markers and echocardiographic indexes in atrial fibrillation (AF) | Baseline
  1. Evaluation of the oscillometric technique of an electronic device in blood pressure measurement.
  2. Evaluation of the relationship of blood pressure levels with serum markers and ultrasonographic cardiac indexes.
  3. Evaluation of a 24h ambulatory blood pressure monitoring device (Microlife WatchBPO3) in terms of its diagnostic value for the detection of atrial fibrillation compared with the reference 24h Holter ECG

CONTACTS AND LOCATIONS:
Overall Officials: George S Stergiou, MD, Study Chair — Hypertension Center,Third Department of Medicine,University of Athens,Greece
Locations (1):
- Hypertension Center, Third Internal Medicine Dpt, University of Athens, Athens, Greece